CLINICAL TRIAL: NCT02228824
Title: The Effect of Very-Low Nicotine Cigarettes on Smoking in Non-Daily Smokers
Brief Title: Very-Low Nicotine Cigarettes and Non-Daily Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saul Shiffman (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Saul Shiffman, Research Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3P30CA047904-25S4 (NIH)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Smoking
Keywords: Smoking; Non-daily smokers; Ecological Momentary Assessment; Biomarkers
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Very low nicotine content cigarettes (Experimental)
  Interventions: Drug: Very low nicotine content cigarettes
- Normal nicotine content cigarettes (Active Comparator)
  Interventions: Drug: Normal nicotine content cigarettes

INTERVENTIONS:
Drug: Very low nicotine content cigarettes — 0.07 mg nicotine delivery
  Arms: Very low nicotine content cigarettes
Drug: Normal nicotine content cigarettes — 0.8 mg nicotine delivery
  Arms: Normal nicotine content cigarettes

SUMMARY:
The purpose of this research study is to investigate the impact of different nicotine levels in cigarettes among non-daily smokers. This research may help inform the Food and Drug Administration (FDA) on how best to regulate tobacco products in the future, with the goal of improving public health.

DETAILED DESCRIPTION:
The overall goal of the study is to assess the effects of switching to Very-Low-Nicotine-Content cigarettes (VLNCCs) among non-daily, or intermittent smokers (ITS). This is a two-arm randomized study with an own-cigarette baseline control. After a 2-week baseline period smoking their own cigarettes, 455 ITS will be randomized (double-blind) for 10 weeks to smoke experimental cigarettes, either: (a) normal nicotine content cigarettes (NNCCs; 0.8 mg) or (b) VLNCCs (0.07 mg), each matched to menthol status of subjects' preferred brand. ITS are more likely to be African-American (AA) smokers; thus AA smokers will be oversampled (to one third of the total sample). Change in cigarette consumption is the primary end-point, and biomarkers of smoke exposure and measures of smoking intensity are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, and smoking cigarettes for at least 3 years
* smoking, on average, 4-27 days per month
* smoking at current rate for at least the previous 3 months
* willingness to try novel cigarettes

Exclusion Criteria:

* active plans to quit or actively seeking smoking cessation treatment in the next 3 months
* severe psychiatric disorders that may interfere with study procedures
* current, regular (i.e., monthly or more) use of nicotine replacement or other tobacco products, by self-report
* exclusive use of roll-your-own cigarettes (since the study uses manufactured cigarettes)
* [for female participants] being pregnant or breastfeeding, or planning to become pregnant, by self-report
* current use of medications such as Chantix (varenicline), Zyban, Wellbutrin, or bupropion for any purpose, including stopping smoking
* occurrence of heart attack, stroke, or angina in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul Shiffman, PhD, Principal Investigator — University of Pittsburgh, Department of Psychology
Locations (1):
- Smoking Research Group, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Shiffman S, Kurland BF, Scholl SM, Mao JM. Nondaily Smokers' Changes in Cigarette Consumption With Very Low-Nicotine-Content Cigarettes: A Randomized Double-blind Clinical Trial. JAMA Psychiatry. 2018 Oct 1;75(10):995-1002. doi: 10.1001/jamapsychiatry.2018.1831. PMID 29902305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the greater Pittsburgh area from June 2015 through April 2017 via various channels (e.g., advertisements on local television stations, public transportation, and social media such as Facebook and Instagram), as well as through University-housed research registries and recruiting services.
Pre-assignment Details: Participants may have been excluded from the study after enrollment but before assignment to an arm if they were found to be unable to adhere to the study protocol or were unable to attend study visits, opted to no longer participate, or if they became unable to contact (i.e., were lost to follow-up).
Period: Overall Study
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Started | 118 | 120
Completed | 89 | 98
Not Completed | 29 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 118 | 120 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (13.5) | 38.4 (14.2) | 37.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 71 | 130
  Male | 59 | 49 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 76 | 76 | 152
  Race: Black | 27 | 34 | 61
  Race: Other | 15 | 10 | 25
Region of Enrollment [Number; unit: participants]
  United States | 118 | 120 | 238
Cigarettes per day at enrollment (across all days) [Mean (Standard Deviation); unit: cigarettes per day] — Average cigarettes per day, across all calendar days in the month preceding initial visit, reported via calendar-based TimeLine Follow-Back
  cigarettes per day | 1.9 (1.6) | 1.9 (1.7) | 1.9 (1.7)
Smoking days per week at enrollment [Mean (Standard Deviation); unit: smoking days per week] — Average smoking days per week, across all calendar days in the month preceding initial visit, reported via calendar-based TimeLine Follow-Back
  smoking days per week | 3.7 (1.4) | 3.7 (1.4) | 3.7 (1.4)
Cigarettes per day at enrollment (smoking days only) [Mean (Standard Deviation); unit: cigarettes per day] — Average cigarettes per day (across smoking days only) in the month preceding initial visit, reported via calendar-based TimeLine Follow-Back
  cigarettes per day | 3.3 (2.3) | 3.5 (2.9) | 3.4 (2.6)
Previous history of daily smoking [Count of Participants; unit: Participants] — Those participants who reported having previously smoked daily, continuously for at least six months, were classified as past daily smokers
  Participants | 57 | 61 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in Cigarette Consumption
Description: Difference in mean daily cigarette consumption between initial two-week baseline period and final two weeks of experimental period, using imputed data
Time Frame: Two-week pre-intervention baseline period compared to final two weeks of 10-week intervention period
Population: All participants who were randomized to an experimental condition (either very-low-nicotine-content cigarettes or normal-nicotine-content cigarettes)
Measure: Least Squares Mean (95% Confidence Interval); unit: cigarettes per day
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 118 | 120
cigarettes per day | -1.6 [-2.0 to -1.1] | -0.05 [-0.5 to 0.4]
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA was performed on 25 sets of imputed data and then analyzed using SAS PROC MIANALYZE; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [0.86 to 2.17]

2. Secondary Outcome: Exposure Measure - Solanesol
Description: The concentration of solanesol, a stable marker indicator of how much smoke has passed through the filter of a smoked cigarette to the smoker, will be assayed as a measure of smoking intensity. The filter of a cigarette butts smoked during the baseline period will be compared to those smoked during the experimental period.
Time Frame: Post-randomization time points at study weeks 4, 8, 12
Measure: Least Squares Mean (Standard Error); unit: mg/butt
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 118 | 120
mg/butt | NA (NA) — Data for this measure will not be analyzed due to the inability of the laboratory at which the analysis was to be performed to conduct these assays, as a result of cuts in CDC funding. | NA (NA) — Data for this measure will not be analyzed due to the inability of the laboratory at which the analysis was to be performed to conduct these assays, as a result of cuts in CDC funding.

3. Secondary Outcome: Exposure Measure - Smoking Topography
Description: Difference between average puff volume per cigarette at laboratory smoking topography sessions at study weeks 4, 8, and 12 across all participants, comparing those assigned to the very-low-nicotine-content cigarette condition to those assigned to the normal-nicotine-content cigarette condition. Topography measures were averaged across all time points for each treatment group.
Time Frame: Post-randomization study visits at study weeks 4, 8, 12
Population: Analysis consists of those participants who contributed data to the study through at least study week 4.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 99 | 101
mL | 501.20 (13.5) | 539.70 (12.83)
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Final Values) = -38.50, 95% CI 2-sided [-75.21 to -1.78]

4. Secondary Outcome: Exposure Measure - Cotinine (Logged)
Description: Cotinine nicotine exposure measure, analyzed from urine samples taken at study office visits
  The natural logarithm (ln) of the cotinine measures was used for analysis.
  Difference in ln(cotinine) between baseline and end of study, from imputed data
Time Frame: Post-randomization office visits weeks 2 (end of baseline period) and 12 (end of study)
Measure: Mean (95% Confidence Interval); unit: log ng/mL
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 118 | 120
log ng/mL | -0.84 [-1.29 to -0.39] | -0.15 [-0.49 to 0.18]
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p = 0.016, ANCOVA; ANCOVA was performed on 25 sets of imputed data and then analyzed using SAS PROC MIANALYZE; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.26 to -0.13]

5. Secondary Outcome: Exposure Measure - Cigarette Butt Weight
Description: Mean mass smoked per cigarette (calculated as the starting cigarette weight minus returned butt weight) aggregated for all cigarettes smoked among participants assigned to the very-low-nicotine-content cigarette, compared to those assigned to the normal-nicotine-content cigarette condition.
Time Frame: Entire length of study, through completion, up to 12 weeks
Population: Analysis population consists of those participants who contributed data to the study for (at minimum) the two-week baseline study period block as well as the first two-week block post-randomization
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 111 | 114
grams | 0.58 (0.01) | 0.60 (0.01)
Statistical Analysis 1: Comparison: Very Low Nicotine Content Cigarettes vs Normal Nicotine Content Cigarettes; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.04 to -0.002]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant during the time of enrollment to completion of the study. Enrollment of study participants began in June 2015 and data collection concluded in July 2017. Thus, adverse event data for the entire study was collected over a 26 month span. Each individual participant participated in the study for 12 weeks.
Description: Adverse events were assessed during study visits via in-session interactions in which study participants were prompted to describe their experiences since the prior visit in an open-ended form, as well as via the self-completed Respiratory Health Questionnaire administered to participants at study visits.
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/120
Serious Adverse Events (participants affected / at risk) | 1/118 | 2/120
Other Adverse Events (participants affected / at risk) | 41/118 | 42/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=118) | Normal Nicotine Content Cigarettes (N=120)
Hospitalization for acute change in mental status (tranisient, unknown etiology) (General disorders) | 0 (0) | 1 (1)
Hospitalization for mini-seizures (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization for psychiatric medication management (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Very Low Nicotine Content Cigarettes (N=118) | Normal Nicotine Content Cigarettes (N=120)
Respiratory (cough, cold) (Respiratory, thoracic and mediastinal disorders) | 33 | 30
Nausea / flu (Gastrointestinal disorders) | 2 | 8
Seasonal allergies (Immune system disorders) | 8 | 9
Headache (Nervous system disorders) | 1 | 1
Acid reflux (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02228824/Prot_SAP_000.pdf